CLINICAL TRIAL: NCT05229107
Title: Randomized Controlled Pilot Trial of Cereset Research For Chronic Nausea
Brief Title: Cereset Research For Chronic Nausea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Both Co-PI, Dr. Ken Koch and Dr. Rajeski, have both left the institution, so we have not been able to receive referrals since their departure.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Susanne Marcus Collins Foundation, Inc. (Other); Gastroenterology Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00078418
Record Dates: First submitted 2021-12-28; First posted 2022-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-06

CONDITIONS: Nausea; Gastroparesis; Stress; Anxiety; Hyperarousal; Quality of Life; Vomiting; Heart Rate Variability
Keywords: nausea; gastroparesis; stress; anxiety; insomnia; quality of life; neurotechnology; autonomic dysregulation; hyperarousal; brain electrical activity; acoustic stimulation; HIRREM; Cereset research; water load satiety testing; Electrogastrography
MeSH Terms: conditions — Nausea; Gastroparesis; Anxiety Disorders; Vomiting; Sleep Initiation and Maintenance Disorders; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: This will be a single site, open label, randomized, wait-list controlled, pilot clinical trial. This study will enroll up to 24 adults, age 18 or older, who have symptoms of chronic nausea (due to gastroparesis and who are not taking medications or supplements for management of symptoms) with a goal of 20 to complete the intervention. Participants will be randomly assigned to either an Early Intervention (EI) group which will receive 6 CR sessions over 4 weeks of audible tones echoing current brainwave activity, following enrollment, or a Delayed Intervention (DI) group which will continue current care only and will serve as a control group. Participants in both groups will continue their other current care throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cereset Research (Active Comparator): Intervention arm using 6 CR sessions
  Interventions: Device: Cereset Research
- Continued Current Care (No Intervention): Participants will continue their current care.

INTERVENTIONS:
Device: Cereset Research — Device: Cereset Research The upgraded platform for medical research using the HIRREM technology has been rebranded as Cereset Research® (CR). This system uses the same core technology and algorithms to echo brainwaves in real-time using audible tones, as with HIRREM. The CR system also includes 64-bit processing architecture for faster feedback, the use of 4 sensors, and the use of standard protocols (with flexibility regarding the length and sequencing of the standard protocols), all done with eyes closed. Four sensors are applied to the scalp at a time. However, only two sensors are actively echoing feedback. The software automatically switches from one sensor pair to the other when needed. This reduces the number of sensor placement changes needed, resulting in shorter session time and fewer interruptions.
  Arms: Cereset Research

SUMMARY:
This study will explore the use of Cereset Research for symptoms associated with refractory chronic nausea in patients with gastroparesis (GP) in a randomized, clinical trial.

DETAILED DESCRIPTION:
Cereset Research (CR) is a noninvasive, close-loop, acoustic stimulation brain feedback system. CR translates brainwaves in real time, echoing them immediately via earbuds. This supports the brain to auto calibrate, self adjust, and relax (acoustic neuromodulation). The brain wave patterns are observed to shift towards improved balance and reduced hyperarousal, getting unstuck from what have become stuck patterns related to trauma and stress. Previous clinical trials using CR, as well as the legacy technology HIRREM, have shown significant benefit to reduce symptoms (stress, anxiety, depression, insomnia, Post-traumatic stress disorder (PTSD), persistent post-concussion symptoms, hot flashes, and others). Improved autonomic nervous system function has also been documented) heart rate variability and variable reflex sensitivity), as well as improved network connectivity on functional Magnetic resonance imaging (MRI) before and after the intervention.

Gastroparesis with normal gastric emptying, and associated chronic nausea, is a challenging clinical condition. There is associated autonomic dysfunction, along with many behavioral symptoms, and effective treatments are lacking. Based on prior studies, there is a reason to believe that CR may have beneficial effects for such patients. This controlled clinical trial will enroll up to 24 adults, age 18 or older, who have symptoms of chronic nausea (due to gastroparesis and who are not taking medications or supplements for management of symptoms) with a goal of 20 to complete the intervention. Participants will be randomly assigned to either an Early Intervention (EI) group which will receive 6 CR sessions over 4 weeks of audible tones echoing current brainwave activity, following enrollment, or a Delayed Intervention (DI) group which will continue current care only and will serve as a control group. Participants in both groups will continue their other current care throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic drug- refractory, nausea and vomiting (ages 18 and up)
* Solid-phase gastric emptying studies show either normal gastric emptying or delayed gastric emptying
* Referring physician will confirm eligibility based on Rome-IV criteria
* Normal upper endoscopy or upper GI series and normal gallbladder tests
* Stable gastrointestinal symptoms with total GCSI score of greater than or equal to 21
* Ability to sign informed consent
* Ability to comply with basic instructions and be able to sit still, comfortably during sessions
* Willingness to complete the EGG and WLST

Exclusion Criteria:

* Non-gastrointestinal disorders which could explain symptoms in the opinion of the investigator
* Active H pylori infection
* Significant hepatic injury (elevated ALT, AST, bilirubin)
* Metabolic, mechanical, or mucosal inflammatory causes to explain GI symptoms such as inflammatory bowel disease, celiac disease, liver or pancreatic disease, or bowel obstruction
* Patients with significant cardiac or cardiovascular disease, malignancy, or other comorbid conditions
* Use of narcotics more than three days per week or other drugs that affect motility (that cannot be held)
* Previous diagnosis or history of neurocardiogenic syncope, orthostatic hypotension, etc.
* Patients with pace makers
* Use of beta blockers which can interfere with heart rate variability recording
* Unable, unwilling, or incompetent to provide informed consent/assent
* Physically unable to come to the study visits, or to sit still, comfortably in a chair for up to 1.5 hours
* Severe hearing impairment (because the subject will be using ear buds during CR)
* Anticipated and ongoing use of alcohol or recreational drugs
* Weight is over the chair limit (400 pounds)
* Currently enrolled in another active intervention research study
* Prior use of: HIRREM, HIRREM-SOP, Brainwave Optimization (BWO), Cereset, Cereset Home, or a wearable configuration of the same (B2, or B2v2)
* Prior use of the following modalities within one month before enrollment: electroconvulsive therapy (ECT), prior use of transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), alpha stimulation, eye movement desensitization and reprocessing (EMDR), brain spotting, neurofeedback, biofeedback, or deep brain stimulation (DBS)
* Known seizure disorder or unspecified seizure within the past 12 months
* Thoughts of suicide within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Gastroparesis Cardinal Symptom Index (GCSI) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Gastroparesis Cardinal Symptom Index (GCSI) is a 9-item scale within the Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM).episodes). The severity of symptom response scale ranges from 0 ("none"), 1 ("mild"), 2 ("moderate"), 3 ("severe") to 4 ("very severe").
  Score can range from 0 to 4. High scores reflect greater symptom severity.
Change in Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGY-SYM) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) is 20 items. This inventory includes six subscales of related GI distress including heartburn/regurgitation, fullness/early satiety, nausea/vomiting, bloating, upper abdominal pain, and lower abdominal pain. Individual item scores range from 0 (none) to 5 (very severe). The higher the score, the more severe the GI symptoms.

SECONDARY OUTCOMES:
Change in Nausea Profile (NP) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Nausea Profile evaluates the experience of 3 dimensions which are involved in the complex feeling of nausea; somatic distress, Gastrointestinal (GI) distress, and emotional distress. The degree to which the patient felt/feels each of the following descriptors during the nauseous period is rated by the patient on a scale of 0 (not at all) to 9 (severely). Higher scores suggest more nausea.
Change in Center for Epidemiologic Studies Depression Scale (CES-D) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a depression scale, which will help to assess this co-morbidity. CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off. The higher the score, the more suggestive of depressive symptoms.
Change in Generalized Anxiety Disorder-7 (GAD-7) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Generalized Anxiety Disorder-7 (GAD-7) is a seven-item screening tool for anxiety that is widely used in primary care. GAD-7 is a brief, reliable and valid measure of assessing generalized anxiety disorder. A score of 10 or greater on the GAD-7 represents a reasonable cut point for identifying cases. Cut points of 5, 10, and 15 might be interpreted as representing mild, moderate, and severe levels of anxiety.

OTHER OUTCOMES:
Change in Severity of Insomnia (ISI) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The ISI is a 7 question, self-reported measure to evaluate symptoms of insomnia, with responses from 0-4 for each question, yielding scores ranging from 0-28. Lower scores represent better outcomes.
Change in Post-traumatic stress disorder (PTSD) Checklist for civilians (PCL-C) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The PTSD Checklist for civilians (PCL-C), measures the American Psychiatric Association's Diagnostic and statistical manual of mental disorders (DSM-IV) Criteria B, C, & D of PTSD symptoms based on traumatic life experience either in civilian life. Seventeen items are rated on a Likert scale with a composite score range of 17 to 85. A score of 44 or higher correlates with probability of civilian-related PTSD. Higher scores suggest more traumatic stress.
Change in Perceived Stress Scale (PSS) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Perceived Stress Scale (PSS) is a ten-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale, with answers rated from 0-4, also includes a number of direct queries about current levels of experienced stress. Total scores range from 0-40. A lower score denotes a lower level of perceived stress.
Change in Fatigue Severity Scale (FSS) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  Fatigue Severity Scale (FSS) is a nine-item instrument to assess how fatigue interferes with daily activities. Items are scored on a 7-point scale ranging from 1=strongly disagree to 7=strongly agree. Total scores range from 9 to 63 and the higher the rating demonstrates greater fatigue severity.
Change in Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOl) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) is a specific scale for how Gastrointestinal (GI) symptoms impact quality of life in those with GI disorders. The scale consists of 30-items scored from 0 (none of the time) to 5 (all of the time) with a recall period of the last 2-weeks. Lower scores suggest better outcomes.
Changes in European Quality of Life Five Dimension (EQ-5D) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The self-rating health question from the EQ-5D on a scale of 0-100 (0 = worst imaginable health state, 100 = best imaginable health state) will be administered to get a snapshot of overall health at that point in time.
Change in The Interpersonal Support Evaluation List (ISEL-12) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The Interpersonal Support Evaluation List - Shortened Version (ISEL-12) is a 12-item scale that was modified from a 40-item scale used to assess perceptions of social support. Three dimensions are evaluated: appraisal support, belonging support, and tangible support. Each item is scaled from 1 to 4 for "Definitely True" to "Definitely False." Total scores range from 0-36 and higher scores suggest more social support.
Change in Short Form McGill Pain Questionnaire (MPQ) scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  Short Form McGill Pain Questionnaire (MPQ) will be given to those who also report chronic pain. The MPQ is made up of 78 words and scores range from 0 (no pain) to 78 (severe pain).
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Pain Interference questionnaire scores | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  The PROMIS Short Form Pain Interference questionnaire will be given too those who report chronic pain. The PROMIS short form is a 6-point Likert-type scale, with scores ranging from 1 (had no pain) to 6 (always) over a 7-day recall period. Higher scores suggest more pain interference
Change in Heart Rate Variability (HRV) | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  Measures of heart rate variability in frequency domain will be derived and measures integrated over specified frequency ranges.
Change in Heart Rate (HR) | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  Continuous heart rate will be recorded while participant is breathing normally in seated position for 10 minutes using Faros 180 heart rate monitor (Bittium Corporation, Oulu, Finland). Beat to beat intervals (RRI) files will be generated at 1000 Hz via the data acquisition software. Files will be analyzed with Nevrokard HRV software (by Nevrokard Kiauta, d.o.o., Izola, Slovenia). Recordings will be visually inspected to ensure data quality (dropped beats or gross motion artifacts are excluded) and first 5 minutes of usable tracings will be analyzed.
Change in Baroreflex Sensitivity (BRS) | Baseline to V3 (8-10 weeks following completion of the intervention for EI; Baseline to V5 (8-10 weeks following completion of the intervention for DI)
  BRS calculated by this method is based on quantification of sequences of at least three beats (n) in which SBP consecutively increases (UP sequence) or decreases (DOWN sequence), which are accompanied by changes in the same direction of the RRI of subsequent beats (n+1). The software scans the RRI and SBP records, identifies sequences, and calculates linear correlation between RRI and SBP for each sequence. The mean of all individual regression coefficients (slopes), a measure of sequence BRS, is calculated for Sequence UP, DOWN and ALL (ms/mmHg). Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard BRS software (Nevrokard BRS, Medistar, Ljubljana, Slovenia).
Changes in Healthcare Utilization Survey | V3 (8-10 weeks following completion of the intervention for EI; V5 (8-10 weeks following completion of the intervention for DI)
  Clinic visit counts will be collected (ED, Urgent Care visits).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hale TS, Smalley SL, Walshaw PD, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. Atypical EEG beta asymmetry in adults with ADHD. Neuropsychologia. 2010 Oct;48(12):3532-9. doi: 10.1016/j.neuropsychologia.2010.08.002. Epub 2010 Aug 10. PMID 20705076
- [Background] Hale TS, Smalley SL, Dang J, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. ADHD familial loading and abnormal EEG alpha asymmetry in children with ADHD. J Psychiatr Res. 2010 Jul;44(9):605-15. doi: 10.1016/j.jpsychires.2009.11.012. Epub 2009 Dec 16. PMID 20006344
- [Background] Hale TS, Smalley SL, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. Atypical alpha asymmetry in adults with ADHD. Neuropsychologia. 2009 Aug;47(10):2082-8. doi: 10.1016/j.neuropsychologia.2009.03.021. Epub 2009 Apr 5. PMID 19467358
- [Background] Lazarev VV, Pontes A, Mitrofanov AA, deAzevedo LC. Interhemispheric asymmetry in EEG photic driving coherence in childhood autism. Clin Neurophysiol. 2010 Feb;121(2):145-52. doi: 10.1016/j.clinph.2009.10.010. Epub 2009 Dec 1. PMID 19951847
- [Background] Stroganova TA, Nygren G, Tsetlin MM, Posikera IN, Gillberg C, Elam M, Orekhova EV. Abnormal EEG lateralization in boys with autism. Clin Neurophysiol. 2007 Aug;118(8):1842-54. doi: 10.1016/j.clinph.2007.05.005. Epub 2007 Jun 19. PMID 17581774
- [Background] Thibodeau R, Jorgensen RS, Kim S. Depression, anxiety, and resting frontal EEG asymmetry: a meta-analytic review. J Abnorm Psychol. 2006 Nov;115(4):715-29. doi: 10.1037/0021-843X.115.4.715. PMID 17100529
- [Background] Avram J, Baltes FR, Miclea M, Miu AC. Frontal EEG activation asymmetry reflects cognitive biases in anxiety: evidence from an emotional face Stroop task. Appl Psychophysiol Biofeedback. 2010 Dec;35(4):285-92. doi: 10.1007/s10484-010-9138-6. PMID 20607389
- [Background] Spironelli C, Penolazzi B, Angrilli A. Dysfunctional hemispheric asymmetry of theta and beta EEG activity during linguistic tasks in developmental dyslexia. Biol Psychol. 2008 Feb;77(2):123-31. doi: 10.1016/j.biopsycho.2007.09.009. Epub 2007 Oct 2. PMID 17997211
- [Background] Moscovitch DA, Santesso DL, Miskovic V, McCabe RE, Antony MM, Schmidt LA. Frontal EEG asymmetry and symptom response to cognitive behavioral therapy in patients with social anxiety disorder. Biol Psychol. 2011 Jul;87(3):379-85. doi: 10.1016/j.biopsycho.2011.04.009. Epub 2011 May 13. PMID 21571033
- [Background] Kemp AH, Griffiths K, Felmingham KL, Shankman SA, Drinkenburg W, Arns M, Clark CR, Bryant RA. Disorder specificity despite comorbidity: resting EEG alpha asymmetry in major depressive disorder and post-traumatic stress disorder. Biol Psychol. 2010 Oct;85(2):350-4. doi: 10.1016/j.biopsycho.2010.08.001. Epub 2010 Aug 11. PMID 20708650
- [Background] Rabe S, Beauducel A, Zollner T, Maercker A, Karl A. Regional brain electrical activity in posttraumatic stress disorder after motor vehicle accident. J Abnorm Psychol. 2006 Nov;115(4):687-98. doi: 10.1037/0021-843X.115.4.687. PMID 17100526
- [Background] Metzger LJ, Paige SR, Carson MA, Lasko NB, Paulus LA, Pitman RK, Orr SP. PTSD arousal and depression symptoms associated with increased right-sided parietal EEG asymmetry. J Abnorm Psychol. 2004 May;113(2):324-9. doi: 10.1037/0021-843X.113.2.324. PMID 15122952
- [Background] Marzano C, Ferrara M, Sforza E, De Gennaro L. Quantitative electroencephalogram (EEG) in insomnia: a new window on pathophysiological mechanisms. Curr Pharm Des. 2008;14(32):3446-55. doi: 10.2174/138161208786549326. PMID 19075720
- [Background] Wolynczyk-Gmaj D, Szelenberger W. Waking EEG in primary insomnia. Acta Neurobiol Exp (Wars). 2011;71(3):387-92. doi: 10.55782/ane-2011-1860. PMID 22068747
- [Background] Riemann D, Spiegelhalder K, Feige B, Voderholzer U, Berger M, Perlis M, Nissen C. The hyperarousal model of insomnia: a review of the concept and its evidence. Sleep Med Rev. 2010 Feb;14(1):19-31. doi: 10.1016/j.smrv.2009.04.002. Epub 2009 May 28. PMID 19481481
- [Background] Cohen H, Benjamin J, Geva AB, Matar MA, Kaplan Z, Kotler M. Autonomic dysregulation in panic disorder and in post-traumatic stress disorder: application of power spectrum analysis of heart rate variability at rest and in response to recollection of trauma or panic attacks. Psychiatry Res. 2000 Sep 25;96(1):1-13. doi: 10.1016/s0165-1781(00)00195-5. PMID 10980322
- [Background] Katz-Leurer M, Rotem H, Keren O, Meyer S. Heart rate and heart rate variability at rest and during exercise in boys who suffered a severe traumatic brain injury and typically-developed controls. Brain Inj. 2010 Feb;24(2):110-4. doi: 10.3109/02699050903508234. PMID 20085448
- [Background] Beckham JC, Taft CT, Vrana SR, Feldman ME, Barefoot JC, Moore SD, Mozley SL, Butterfield MI, Calhoun PS. Ambulatory monitoring and physical health report in Vietnam veterans with and without chronic posttraumatic stress disorder. J Trauma Stress. 2003 Aug;16(4):329-35. doi: 10.1023/A:1024457700599. PMID 12895015
- [Background] Spiegelhalder K, Fuchs L, Ladwig J, Kyle SD, Nissen C, Voderholzer U, Feige B, Riemann D. Heart rate and heart rate variability in subjectively reported insomnia. J Sleep Res. 2011 Mar;20(1 Pt 2):137-45. doi: 10.1111/j.1365-2869.2010.00863.x. PMID 20626615
- [Background] Tobaldini E, Nobili L, Strada S, Casali KR, Braghiroli A, Montano N. Heart rate variability in normal and pathological sleep. Front Physiol. 2013 Oct 16;4:294. doi: 10.3389/fphys.2013.00294. PMID 24137133
- [Background] Tsuji H, Larson MG, Venditti FJ Jr, Manders ES, Evans JC, Feldman CL, Levy D. Impact of reduced heart rate variability on risk for cardiac events. The Framingham Heart Study. Circulation. 1996 Dec 1;94(11):2850-5. doi: 10.1161/01.cir.94.11.2850. PMID 8941112
- [Background] Dekker JM, Schouten EG, Klootwijk P, Pool J, Swenne CA, Kromhout D. Heart rate variability from short electrocardiographic recordings predicts mortality from all causes in middle-aged and elderly men. The Zutphen Study. Am J Epidemiol. 1997 May 15;145(10):899-908. doi: 10.1093/oxfordjournals.aje.a009049. PMID 9149661
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Lee EA, Bissett JK, Carter MA, Cowan PA, Pyne JM, Speck PM, Theus SA, Tolley EA. Preliminary findings of the relationship of lower heart rate variability with military sexual trauma and presumed posttraumatic stress disorder. J Trauma Stress. 2013 Apr;26(2):249-56. doi: 10.1002/jts.21797. PMID 23568414
- [Background] Shah AJ, Lampert R, Goldberg J, Veledar E, Bremner JD, Vaccarino V. Posttraumatic stress disorder and impaired autonomic modulation in male twins. Biol Psychiatry. 2013 Jun 1;73(11):1103-10. doi: 10.1016/j.biopsych.2013.01.019. Epub 2013 Feb 21. PMID 23434412
- [Background] Minassian A, Geyer MA, Baker DG, Nievergelt CM, O'Connor DT, Risbrough VB; Marine Resiliency Study Team. Heart rate variability characteristics in a large group of active-duty marines and relationship to posttraumatic stress. Psychosom Med. 2014 May;76(4):292-301. doi: 10.1097/PSY.0000000000000056. PMID 24804881
- [Background] Park J, Marvar PJ, Liao P, Kankam ML, Norrholm SD, Downey RM, McCullough SA, Le NA, Rothbaum BO. Baroreflex dysfunction and augmented sympathetic nerve responses during mental stress in veterans with post-traumatic stress disorder. J Physiol. 2017 Jul 15;595(14):4893-4908. doi: 10.1113/JP274269. Epub 2017 Jun 14. PMID 28503726
- [Background] Park JE, Lee JY, Kang SH, Choi JH, Kim TY, So HS, Yoon IY. Heart rate variability of chronic posttraumatic stress disorder in the Korean veterans. Psychiatry Res. 2017 Sep;255:72-77. doi: 10.1016/j.psychres.2017.05.011. Epub 2017 May 9. PMID 28528244
- [Background] Minassian A, Maihofer AX, Baker DG, Nievergelt CM, Geyer MA, Risbrough VB; Marine Resiliency Study Team. Association of Predeployment Heart Rate Variability With Risk of Postdeployment Posttraumatic Stress Disorder in Active-Duty Marines. JAMA Psychiatry. 2015 Oct;72(10):979-86. doi: 10.1001/jamapsychiatry.2015.0922. PMID 26353072
- [Background] Pyne JM, Constans JI, Wiederhold MD, Gibson DP, Kimbrell T, Kramer TL, Pitcock JA, Han X, Williams DK, Chartrand D, Gevirtz RN, Spira J, Wiederhold BK, McCraty R, McCune TR. Heart rate variability: Pre-deployment predictor of post-deployment PTSD symptoms. Biol Psychol. 2016 Dec;121(Pt A):91-98. doi: 10.1016/j.biopsycho.2016.10.008. Epub 2016 Oct 20. PMID 27773678
- [Background] Kleiger RE, Miller JP, Bigger JT Jr, Moss AJ. Decreased heart rate variability and its association with increased mortality after acute myocardial infarction. Am J Cardiol. 1987 Feb 1;59(4):256-62. doi: 10.1016/0002-9149(87)90795-8. PMID 3812275
- [Background] Carnethon MR, Golden SH, Folsom AR, Haskell W, Liao D. Prospective investigation of autonomic nervous system function and the development of type 2 diabetes: the Atherosclerosis Risk In Communities study, 1987-1998. Circulation. 2003 May 6;107(17):2190-5. doi: 10.1161/01.CIR.0000066324.74807.95. Epub 2003 Apr 14. PMID 12695289
- [Background] Chandra P, Sands RL, Gillespie BW, Levin NW, Kotanko P, Kiser M, Finkelstein F, Hinderliter A, Pop-Busui R, Rajagopalan S, Saran R. Predictors of heart rate variability and its prognostic significance in chronic kidney disease. Nephrol Dial Transplant. 2012 Feb;27(2):700-9. doi: 10.1093/ndt/gfr340. Epub 2011 Sep 12. PMID 21765187
- [Background] Marsac J. [Heart rate variability: a cardiometabolic risk marker with public health implications]. Bull Acad Natl Med. 2013 Jan;197(1):175-86. French. PMID 24672989
- [Background] Thayer JF, Hansen AL, Saus-Rose E, Johnsen BH. Heart rate variability, prefrontal neural function, and cognitive performance: the neurovisceral integration perspective on self-regulation, adaptation, and health. Ann Behav Med. 2009 Apr;37(2):141-53. doi: 10.1007/s12160-009-9101-z. Epub 2009 May 8. PMID 19424767
- [Background] Nolan RP, Jong P, Barry-Bianchi SM, Tanaka TH, Floras JS. Effects of drug, biobehavioral and exercise therapies on heart rate variability in coronary artery disease: a systematic review. Eur J Cardiovasc Prev Rehabil. 2008 Aug;15(4):386-96. doi: 10.1097/HJR.0b013e3283030a97. PMID 18677161
- [Background] Lee SW, Gerdes L, Tegeler CL, Shaltout HA, Tegeler CH. A bihemispheric autonomic model for traumatic stress effects on health and behavior. Front Psychol. 2014 Aug 1;5:843. doi: 10.3389/fpsyg.2014.00843. eCollection 2014. PMID 25136325
- [Background] Bellesi M, Riedner BA, Garcia-Molina GN, Cirelli C, Tononi G. Enhancement of sleep slow waves: underlying mechanisms and practical consequences. Front Syst Neurosci. 2014 Oct 28;8:208. doi: 10.3389/fnsys.2014.00208. eCollection 2014. PMID 25389394
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Background] Sterling P. Allostasis: a model of predictive regulation. Physiol Behav. 2012 Apr 12;106(1):5-15. doi: 10.1016/j.physbeh.2011.06.004. Epub 2011 Jun 12. PMID 21684297
- [Background] Tegeler CH, Kumar SR, Conklin D, Lee SW, Gerdes L, Turner DP, Tegeler CL, C Fidali B, Houle TT. Open label, randomized, crossover pilot trial of high-resolution, relational, resonance-based, electroencephalic mirroring to relieve insomnia. Brain Behav. 2012 Nov;2(6):814-24. doi: 10.1002/brb3.101. Epub 2012 Oct 28. PMID 23170244
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Pajewski NM. Reduction in menopause-related symptoms associated with use of a noninvasive neurotechnology for autocalibration of neural oscillations. Menopause. 2015 Jun;22(6):650-5. doi: 10.1097/GME.0000000000000422. PMID 25668305
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Gerdes L, Shaltout HA, Miles CM, Simpson SL. A Preliminary Study of the Effectiveness of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology in the Treatment of Athletes with Persisting Post-concussion Symptoms. Sports Med Open. 2016 Dec;2(1):39. doi: 10.1186/s40798-016-0063-y. Epub 2016 Sep 14. PMID 27747793
- [Background] Tegeler CL, Gerdes L, Shaltout HA, Cook JF, Simpson SL, Lee SW, Tegeler CH. Successful use of closed-loop allostatic neurotechnology for post-traumatic stress symptoms in military personnel: self-reported and autonomic improvements. Mil Med Res. 2017 Dec 22;4(1):38. doi: 10.1186/s40779-017-0147-0. PMID 29502530
- [Background] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Background] Tegeler CH, Shaltout HA, Tegeler CL, Gerdes L, Lee SW. Rightward dominance in temporal high-frequency electrical asymmetry corresponds to higher resting heart rate and lower baroreflex sensitivity in a heterogeneous population. Brain Behav. 2015 Jun;5(6):e00343. doi: 10.1002/brb3.343. Epub 2015 May 1. PMID 26085968
- [Background] Lee SW, Laurienti PJ, Burdette JH, Tegeler CL, Morgan AR, Simpson SL, Gerdes L, Tegeler CH. Functional Brain Network Changes Following Use of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology for Military-Related Traumatic Stress. J Neuroimaging. 2019 Jan;29(1):70-78. doi: 10.1111/jon.12571. Epub 2018 Oct 10. PMID 30302866
- [Background] Tegeler CL, Howard LJ, Schmidt KD, Cook JF, Kumar S, Simpson SL, Lee SW, Gerdes L, Tegeler CH. 0389 USE OF A CLOSED-LOOP ACOUSTIC STIMULATION NEUROTECHNOLOGY IMPROVES SYMPTOMS OF MODERATE TO SEVERE INSOMNIA: RESULTS OF A PLACEBO-CONTROLLED TRIAL. Sleep. 2017;40:A145-A.
- [Background] Shaltout HA, Tegeler CL, Lee SW, Tegeler CH. 0363 IN SUBJECTS WITH INSOMNIA, USE OF A CLOSED-LOOP ACOUSTIC STIMULATION NEUROTECHNOLOGY IMPROVES HEART RATE VARIABILITY AND BAROREFLEX SENSITIVITY: RESULTS OF A PLACEBO-CONTROLLED CLINICAL TRIAL. Sleep. 2017;40:A135-A
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Kaplan NM RB. Technique of blood pressure measurement in the diagnosis of hypertension. UpToDate. Barkris GL, Sheridan AM, eds. Waltham, MA; 2010.
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Radloff LS. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1977;1:385-401.
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] FW W, BT L, DS H, JA H, TM K. The PTSD Checklist (PCL): Reliability, validity, and diagnostic utility. 9th Annual Meeting of the International Society for Traumatic Stress Studies. San Antonio, TX.
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Offenbacher M, Sauer S, Kohls N, Waltz M, Schoeps P. Quality of life in patients with fibromyalgia: validation and psychometric properties of the German Quality of Life Scale (QOLS-G). Rheumatol Int. 2012 Oct;32(10):3243-52. doi: 10.1007/s00296-011-2184-4. Epub 2011 Oct 30. PMID 22038277
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Bradley KA, DeBenedetti AF, Volk RJ, Williams EC, Frank D, Kivlahan DR. AUDIT-C as a brief screen for alcohol misuse in primary care. Alcohol Clin Exp Res. 2007 Jul;31(7):1208-17. doi: 10.1111/j.1530-0277.2007.00403.x. Epub 2007 Apr 19. PMID 17451397
- [Background] Bradley KA, Bush KR, Epler AJ, Dobie DJ, Davis TM, Sporleder JL, Maynard C, Burman ML, Kivlahan DR. Two brief alcohol-screening tests From the Alcohol Use Disorders Identification Test (AUDIT): validation in a female Veterans Affairs patient population. Arch Intern Med. 2003 Apr 14;163(7):821-9. doi: 10.1001/archinte.163.7.821. PMID 12695273
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] De La Loge C, Trudeau E, Marquis P, Revicki DA, Rentz AM, Stanghellini V, Talley NJ, Kahrilas P, Tack J, Dubois D. Responsiveness and interpretation of a quality of life questionnaire specific to upper gastrointestinal disorders. Clin Gastroenterol Hepatol. 2004 Sep;2(9):778-86. doi: 10.1016/s1542-3565(04)00349-0. PMID 15354278
- [Background] de la Loge C, Trudeau E, Marquis P, Kahrilas P, Stanghellini V, Talley NJ, Tack J, Revicki DA, Rentz AM, Dubois D. Cross-cultural development and validation of a patient self-administered questionnaire to assess quality of life in upper gastrointestinal disorders: the PAGI-QOL. Qual Life Res. 2004 Dec;13(10):1751-62. doi: 10.1007/s11136-004-8751-3. PMID 15651545
- [Background] Cucchiara S, Minella R, Riezzo G, Vallone G, Vallone P, Castellone F, Auricchio S. Reversal of gastric electrical dysrhythmias by cisapride in children with functional dyspepsia. Report of three cases. Dig Dis Sci. 1992 Jul;37(7):1136-40. doi: 10.1007/BF01300300. PMID 1618063
- [Background] Lacy BE, Crowell MD, Mathis C, Bauer D, Heinberg LJ. Gastroparesis: Quality of Life and Health Care Utilization. J Clin Gastroenterol. 2018 Jan;52(1):20-24. doi: 10.1097/MCG.0000000000000728. PMID 27775961
- [Background] Muth ER, Stern RM, Thayer JF, Koch KL. Assessment of the multiple dimensions of nausea: the Nausea Profile (NP). J Psychosom Res. 1996 May;40(5):511-20. doi: 10.1016/0022-3999(95)00638-9. PMID 8803860